CLINICAL TRIAL: NCT06656507
Title: Comparison of the Efficacy of Quadro Iliac Plane Block and Erector Spinae Plane Block on Postoperative Pain Management and Opioid Consumption in Single Level Lumbar Discectomies: A Multicenter Randomized Controlled Trial
Brief Title: Comparison of Quadro Iliac vs Erector Spinae Plane Block on Postoperative Pain and Opioid Use in Lumbar Discectomies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Engin Ihsan Turan, anesthesiology and reanimation specialist, Kanuni Sultan Suleyman Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: qip-esp/ldh
Record Dates: First submitted 2024-10-22; First posted 2024-10-24 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Postoperative Pain; Lumbar Disc Herniation
MeSH Terms: conditions — Pain, Postoperative; Intervertebral Disc Displacement

STUDY DESIGN:
Intervention Model Description: This study follows a Parallel Assignment model where eligible patients undergoing lumbar vertebra surgeries will be randomized into one of two groups. One group will receive the Quadro Iliac Plane Block (QIPB), while the other group will receive the Erector Spinae Plane (ESP) Block. Both interventions will be administered pre-awakening following surgery, with each group receiving only their assigned block. The groups will be assessed independently for postoperative pain control, opioid consumption, side effects, and overall patient satisfaction. This parallel approach ensures that each group's treatment and outcomes are evaluated without crossover, allowing for a direct comparison of the two regional anesthesia techniques.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: This study employs a Double-Blind masking approach to minimize bias. Both the patients and the healthcare providers (including postoperative care staff) will be unaware of which block (Quadro Iliac Plane Block or Erector Spinae Plane Block) was administered. The anesthesiologists performing the blocks will be informed of the assigned intervention but will not participate in postoperative care or outcome assessment. The outcome assessors, who will evaluate pain scores, opioid consumption, and other outcomes, will also be blinded to the group allocation to ensure unbiased data collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Quadro Iliac Plane Block (QIPB) Arm (Experimental): Patients in this arm will receive the Quadro Iliac Plane Block (QIPB) before awakening from lumbar vertebra surgery. Patients in this arm will receive the Quadro Iliac Plane Block (QIPB) before awakening from lumbar vertebra surgery. The patient will be placed in a prone position, and a low-frequency convex ultrasound transducer (2-6 MHz) will be used. The transducer will be placed in the midline at the L3 level in the transverse plane to identify the spinal process. After lateral movement, the transverse process within the erector spinae muscle will be visualized. The transducer will then be rotated to the parasagittal plane and moved caudally to identify the attachment of the Quadratus Lumborum Muscle (QLM) to the iliac crest. A 22G x 100 mm peripheral nerve block needle (Stimuplex® Ultra 360®, B-Braun, USA) will be advanced under ultrasound guidance, and 50 mg (0.25%) bupivacaine will be injected bilaterally into the fascia below the QLM.
  Interventions: Procedure: Quadro Iliac Plane Block (QIPB)
- Erector Spinae Plane Block (ESP) Arm (Experimental): Patients in this arm will receive the Erector Spinae Plane Block (ESP) before awakening from lumbar vertebra surgery. Patients in this arm will receive the Erector Spinae Plane Block (ESP) before awakening from lumbar vertebra surgery. A linear ultrasound probe will be placed transversely over the L3 vertebra to visualize the transverse process. A block needle (Stimuplex® Ultra 360®, B-Braun, USA) will be advanced under ultrasound guidance until it contacts the transverse process. After withdrawing the needle by 1 mm, 50 mg (0.25%) bupivacaine will be injected bilaterally.
  Interventions: Procedure: Erector Spinae Plane Block (ESP)

INTERVENTIONS:
Procedure: Quadro Iliac Plane Block (QIPB) — The Quadro Iliac Plane Block (QIPB) will be performed pre-awakening in patients undergoing lumbar vertebra surgeries. Using a low-frequency convex ultrasound transducer (2-6 MHz), the spinal process will be identified at the L3 level in a prone-positioned patient. The transducer will be moved laterally to locate the transverse process within the erector spinae muscle and then rotated to the parasagittal plane to identify the Quadratus Lumborum Muscle (QLM) attachment to the iliac crest. A 22G x 100 mm block needle will be advanced under ultrasound guidance, and 50 mg (0.25%) bupivacaine will be injected bilaterally into the fascia beneath the QLM. This technique is designed to provide effective postoperative pain control by blocking the nerves in the quadratus lumborum plane.
  Arms: Quadro Iliac Plane Block (QIPB) Arm
Procedure: Erector Spinae Plane Block (ESP) — The Erector Spinae Plane Block (ESP) will also be performed pre-awakening. A linear ultrasound probe will be placed transversely at the level of the L3 vertebra to visualize the transverse process. A block needle will be advanced under ultrasound guidance until it touches the transverse process, after which the needle will be withdrawn 1 mm. Fifty milligrams (0.25%) bupivacaine will then be administered bilaterally. The ESP block aims to provide postoperative analgesia by blocking sensory nerves in the erector spinae plane.
  Arms: Erector Spinae Plane Block (ESP) Arm

SUMMARY:
This multicenter, randomized, controlled study aims to compare the analgesic efficacy of Quadro Iliac Plane Block (QIPB) and Erector Spinae Plane (ESP) Block in lumbar vertebra surgeries. The study will evaluate postoperative pain management, opioid consumption, side effects, hospital stay duration, and patient satisfaction. Patients scheduled for single-level lumbar disk herniation surgery will be randomized to receive either the QIPB or ESP block before awakening from anesthesia. Pain scores will be measured at multiple postoperative time points, and opioid consumption will be monitored using patient-controlled analgesia (PCA). The study seeks to identify the most effective and safe method for postoperative pain management in lumbar surgeries.

DETAILED DESCRIPTION:
Detailed Description: The purpose of this study is to compare the analgesic efficacy of two commonly used regional anesthesia techniques-Quadro Iliac Plane Block (QIPB) and Erector Spinae Plane (ESP) Block-in lumbar vertebra surgeries. This is a prospective, randomized, controlled, and multicenter trial. The study aims to evaluate the effectiveness of QIPB and ESP blocks in postoperative pain control, opioid consumption, side effects, hospital stay duration, and patient satisfaction. The findings are expected to contribute to identifying more effective and safer methods for postoperative pain management in lumbar spine surgeries.

This study will focus on examining the impact of these two different block techniques on pain scores, particularly during the early postoperative period. By analyzing the potential benefits and limitations of these techniques, the study will aim to provide valuable insights into postoperative pain control. Additionally, a comparative analysis of the feasibility and patient safety of both block techniques will be conducted.

Materials and Methods: Patients aged 18 and above, with ASA scores of I-III, without bleeding diathesis, no history of anticoagulant use, no history of allergies to the medications used, and no history of neuropathic disease, undergoing single-level lumbar disk herniation surgery will be included in the study. Patients will be randomized to receive either ESP or QIP block before awakening post-surgery. Informed consent will be obtained from all participants, and both blocks will be thoroughly explained.

To avoid bias, the study is designed as multicenter, and experienced anesthesiologists will perform the blocks at the end of the surgery, before the patient is awakened.

Block Techniques:

ESP Block: With a linear ultrasound probe in the transverse plane, the transverse process of the L3 vertebra will be identified. A block needle will be advanced under ultrasound guidance, and once the needle touches the transverse process, it will be withdrawn by 1mm, confirmed with sterile saline, and 50 mg (0.25%) bupivacaine will be administered bilaterally.

QIP Block: For patients in a prone position, a low-frequency convex transducer (2-6 MHz) will be placed at the midline at the L3 level in the transverse plane to identify the spinal process. Lateral movement will identify the transverse process within the erector spinae muscle. The transducer will then be rotated to the parasagittal plane and moved caudally to locate the attachment of the Quadratus Lumborum Muscle (QLM) to the iliac crest. A block needle will be advanced under ultrasound guidance, and 50 mg (0.25%) bupivacaine will be injected bilaterally into the fascia below the QLM.

Postoperative Care: Before awakening, all patients will receive 1g of paracetamol, 100mg of tramadol, and 50mg of dexketoprofen intravenously. Postoperatively, multimodal analgesia will be provided using patient-controlled analgesia (PCA) with tramadol HCl, set to deliver 20 mg boluses with a lockout interval of 20 minutes, and a maximum dose limit of 200mg over 4 hours. Pain scores will be assessed at rest and with movement at 0, 2, 6, 12, and 24 hours using the Numeric Rating Scale (NRS), ranging from 0-10. Opioid consumption and the need for rescue analgesia (50 mg dexketoprofen in 100cc saline over 20 minutes) will also be evaluated. Routine administration of 1g of intravenous paracetamol will be given at 6 hours postoperatively.

Sample Size and Statistical Methods: A power analysis with an alpha error of 0.05, power of 0.8, and effect size of 0.8 determined that at least 26 patients per group (total 52) are needed. Accounting for potential errors, 60 patients will be enrolled in the study. Data will be analyzed using IBM SPSS 21. Descriptive statistics will be computed for each variable, with continuous data presented as mean ± standard deviation or median (IQR), and categorical data as frequencies and percentages. The Shapiro-Wilk test will be used to assess normality, and non-parametric tests will be applied if the data are not normally distributed.

Between-group comparisons of continuous data will use independent t-tests or Mann-Whitney U tests, depending on normality. Categorical variables will be compared using the Chi-square test or Fisher's Exact Test. Primary outcomes, including NRS pain scores at rest at 24 hours, will be analyzed using t-tests or Mann-Whitney U tests. Secondary outcomes, such as opioid consumption, nausea, vomiting, and motor block, will be analyzed similarly. Rescue analgesia need will be analyzed with the Chi-square test. A p-value of <0.05 will be considered statistically significant.

This study aims to provide crucial information on the efficacy and safety of both block techniques, potentially improving postoperative pain management practices in lumbar spine surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 65 years.
* ASA physical status classification I-III.
* Patients scheduled for single-level lumbar disk herniation surgery.
* No history of bleeding diathesis.
* No history of anticoagulant use.
* No known allergies to the medications used in the study (e.g., bupivacaine).
* No history of neuropathic diseases.
* Patients who have provided informed consent to participate in the study.

Exclusion Criteria:

* Patients younger than 18 or older than 65 years.
* ASA physical status classification IV or higher.
* Patients with a history of coagulopathy or bleeding disorders.
* Patients with a history of chronic opioid use or substance abuse.
* Patients with allergies to local anesthetics (e.g., bupivacaine).
* Patients with significant neuropathic conditions or central nervous system disorders.
* Patients with any contraindication to regional anesthesia.
* Pregnant or breastfeeding women.
* Patients unable to provide informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-16 (Actual)

PRIMARY OUTCOMES:
NRS Score | 24 hours
  Postoperative pain assessed by numerical rating scale (NRS) (0-10)

SECONDARY OUTCOMES:
PCA | 24 hours
  PCA(patient controlled analgesia) opioid consumption
Rescue analgesia | 24 hours
  Number of participant need rescue analgesia requirement (deksketoprofen 50mg)
Side effects | 24 hours
  Side effects (nausea, vomiting, motor block)

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Health Science University İstanbul Kanuni Sultan Süleyman Education and Training Hospital, Istanbul
  - Zincirlikuyu Medicana Hospital, Istanbul

IPD SHARING:
Plan to Share IPD: Undecided